CLINICAL TRIAL: NCT03447756
Title: A Randomized, Placebo-Controlled, Optimized Titration Study of ABX-1431 in Adult Patients With Peripheral Neuropathic Pain
Brief Title: Titration Study of ABX-1431
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Abide Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ABX-1431_PN014
Record Dates: First submitted 2018-02-09; First posted 2018-02-27 (Actual); Last update posted 2019-07-12 (Actual); Status verified 2019-07

CONDITIONS: Post Herpetic Neuralgia; Diabetic Peripheral Neuropathy; Small Fiber Neuropathy; Post-Traumatic Neuralgia
MeSH Terms: conditions — Neuralgia, Postherpetic; Small Fiber Neuropathy | interventions — ABX-1431

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ABX-1431 (Experimental): One or more oral capsules containing 2 mg or 10 mg or 50 mg of ABX-1431 HCl or matching placebo are administered daily to enrolled patients. Patients will undergo a blinded dose escalation. All patients will receive placebo on some days to assess safety and neuropathic pain. Patients will undergo an optimized titration of ABX-1431 HCl with the daily dose between 8 mg and 24 mg of ABX-1431. Each patients dose will be determined by the Investigator based on assessment of adverse events.
  Interventions: Drug: ABX-1431
- Placebo oral capsule (Placebo Comparator): One or more oral capsules containing placebo are administered daily to enrolled patients. Patients will undergo a blinded dose escalation. All patients will receive placebo on some days to assess safety and neuropathic pain. Patients will undergo an optimized titration of placebo. Each patients dose will be determined by the Investigator based on assessment of adverse events.
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Drug: ABX-1431 — Capsules of either 2mg, 10mg, or 50mg
  Arms: ABX-1431
Drug: Placebo oral capsule — placebo to match
  Arms: Placebo oral capsule

SUMMARY:
This study is designed to identify a titration regimen of ABX-1431 in adults with neuropathic pain with satisfactory tolerability to central nervous system (CNS) adverse events (AEs). During the course of this study, each participant will take a daily dose of ABX-1431 or a matching placebo for 28 days.

DETAILED DESCRIPTION:
This is a double-blind, placebo-controlled, optimized titration study of ABX-1431 HCl. The study will explore whether patients experiencing ABX-1431-related CNS AE accommodate or become tolerant to them with continued dosing. The efficacy of ABX-1431 in treating neuropathic pain will be assessed by the change from baseline in pain intensity scores using numerical rating scale (NRS-11).

All patients will undergo a screening visit for enrollment criteria. Eligible patients will be treated with daily medication for 28 days which will include some treatment with placebo and some treatment with ABX-1431 HCl. Patients will record their daily average pain using a paper numerical rating scale (NRS-11).

This study will enroll up to 32 patients with peripheral neuropathic pain due to one of the four following diagnostic groups: post-herpetic neuralgia, diabetic peripheral neuropathy, small fiber neuropathy or post-traumatic neuropathic pain.

ELIGIBILITY:
Key Inclusion Criteria:

* Patient is a male or female over the age of 18 years of age at the Screening Visit.
* Patient has a peripheral neuropathic pain in one of the following diagnostic groups that is persistent for > 3 months

  * Post-herpetic neuralgia
  * Diabetic peripheral neuropathy
  * Small fiber neuropathy
  * Post-traumatic neuropathic pain
* Patient's median NRS-11 pain intensity score must be ≥ 4 during the baseline period
* If a patient enters the trial on daily background neuropathic pain medications, then the patient must be on stable dose of medications for at least 30 days before enrollment and throughout the study.
* Patient is able to understand and comply with the protocol procedures for the entire trial and must give written informed consent.
* Men and Women must agree to a medically approved contraceptive regimen.

Key Exclusion Criteria:

* Patient is taking potent cytochrome P450 3A4/5 inducers or inhibitors
* Patient has received injection therapies (e.g., botulinum toxin, anesthetic or nerve block) or transcutaneous electrical stimulation to control pain in the past 60 days
* Patient has evidence of alcohol, drug or chemical abuse in the year before the Screening Visit.
* Patient is a lactating or pregnant female or a female who intends to become pregnant within 90 days following the last dose of investigational product.
* Patient has specific laboratory abnormalities

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2017-10-02 (Actual); Primary Completion 2019-05-07 (Actual); Study Completion 2019-05-07 (Actual)

PRIMARY OUTCOMES:
Identify a titration regimen of ABX-1431 | 28 days
  The number of patients unable to continue due to central nervous system (CNS) adverse events (AEs) while exceeding mean plasma ABX-1431 AUC_0-24 of 190 ng*hr/ml or inhibiting 2-arachidonoylglycerol (2-AG) hydrolysis in peripheral blood mononuclear cells (PBMC) by more than 62% time-weighted inhibition over 24-hours.

SECONDARY OUTCOMES:
Tolerance to ABX-1431 related CNS AEs determined by whether or not AEs resolve with continued dosing | 28 days
Numerical Rating Scale (NRS-11) | 20 days
  Change from Baseline in Pain Scores on the Numerical Rating Scale-11 (NRS-11) at 20 days.

CONTACTS AND LOCATIONS:
Overall Officials: Vitale Lisnic, PhD, Principal Investigator — ARENSIA EXPLORATORY MEDICINE
Locations (1):
- Republican Clinical Hospital, Chisinau, Moldova

IPD SHARING:
Plan to Share IPD: No